CLINICAL TRIAL: NCT05297019
Title: Hyperbaric Dosage Analysis Effect Of Various PO2 Exposures: Hyperoxia-Hypoxia Paradox On Stem Cell Mobilization, Cell Signaling, Inflammation, Epigenetics & Cell Regeneration
Brief Title: A Dosing Study of Hyperbaric Oxygen Therapy (HBOT) on Epigenetic Aging
Acronym: HBOT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: TruDiagnostic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: SM-TD-001
Record Dates: First submitted 2022-03-04; First posted 2022-03-25 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Aging
MeSH Terms: interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: The "control" group will crossover to active treatment after 3 months of observation.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, the principal investigator, and outcomes assessor will be blinded to patient's HBOT dosing. Technicians at the clinic will know which treatment dose each participant is receiving in order to deliver appropriate dosing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Mild pressure HBOT (Experimental): "Mild" pressure HBOT: 100% O2 @ 4.2 PSI for 100 minutes 3x/week for 6 weeks, 2 weeks off, and then an additional 4 weeks of therapy. Followed by 3 months of no treatment
  Interventions: Procedure: Hyperbaric Oxygen Therapy
- Arm 2: High pressure HBOT (Experimental): "High" pressure HBOT: 100% O2 @ 14 PSI for 100 minutes 3x/week for 6 weeks, 2 weeks off, and then an additional 4 weeks of therapy. Followed by 3 months of no treatment
  Interventions: Procedure: Hyperbaric Oxygen Therapy
- Arm 3: Crossover Arm (Experimental): Patients will have 3 months of no treatment, and then be randomized to receive either high pressure or mild pressure HBOT
  Interventions: Procedure: Hyperbaric Oxygen Therapy

INTERVENTIONS:
Procedure: Hyperbaric Oxygen Therapy — hyperbaric oxygen therapy

SUMMARY:
This study aims to assess the impact of hyperbaric oxygen therapy on a number of outcomes, including epigenetic aging, inflammation, and cellular health.

DETAILED DESCRIPTION:
While current research has identified many mechanisms of action, effects and cell signaling benefits resulting from HBOT, we do not have a firm understanding of the timeframe and dosage for many of these expected adaptations. Data from this study will be collected and shared on an ongoing basis throughout the course of care. This research project will help us to confirm these cell-signaling changes and benefits, and also develop a better understanding of the necessary PO2 and time frame required in order to achieve these changes leading to improved patient outcomes in the field of hyperbaric medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Any sex, gender orientation, and ethnicity
2. Between ages 40 and 70
3. Must be willing and able to participate in venipuncture, health history and clinical assessments, lab test assessment, hyperbaric oxygen treatment.
4. Participants must also agree to maintain their current lifestyle choices consistent with pre- participation with this study. Participants should not change their exercise programs, diets, sleep patterns supplements or other. Any significant changes in their lifestyle choices must be reported to the staff.

Exclusion Criteria:

1. Significant change in diagnosis and/or treatment of major illness or injury within 2 years prior to screening, e.g., diabetes, cancer, cardiovascular disease, psychiatric condition
2. Any ongoing immune system concerns or immunodeficiency disease
3. Body mass index (BMI) changes of more than 5% over the course of the study
4. Changes in weight of more than 15 lbs. during the course of the study
5. Presence of a severe active infection as determined by the principal investigator.
6. Any other illness, disorder, alcohol or chemical dependence that in the opinion of investigators would render study participation unsuitable
7. Unable or unwilling to provide required biological sample
8. Unable or unwilling to avoid pregnancy during study period
9. Presence of cataracts before the study begins
10. Myopic changes within the first 30 days of treatment

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Epigenetic Aging | Testing will compare baseline with 6 months
  DNA methylation of blood samples for epigenetic age

SECONDARY OUTCOMES:
Neurotrax | Testing will compare baseline with 6 months
  Brain Care brain fitness tests follow the neuropsychological tradition by measuring:
  Memory, Executive Function, Attention, Visual Spatial, Verbal Function, Problem Solving, Working Memory. These tests are performed on a computer through a secure online assessment procedure. The scores on these tests are aggregated to create on measure of brain fitness

CONTACTS AND LOCATIONS:
Locations (1):
- New Jersey HBOT, Florham Park, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided